CLINICAL TRIAL: NCT05671484
Title: Investigation of the Effects of Transversalis Fascial Plane Block and Quadratus Lumborum Plane Block Applied in Pediatric Infra-umbilical Surgeries on Postoperative Pain and Analgesic Consumption
Brief Title: TFPB vs QLB III in Infra-umbilical Pediatric Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Onur Baran, Assistant Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.205.11.06
Record Dates: First submitted 2022-12-31; First posted 2023-01-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Transversalis Fascial Plane Block; Quadratus Lumborum Block; Analgesia; Pediatric; Ultrasound Guidance
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into two equal groups.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis Fascial Plane Block Group (Active Comparator): Patients will receive ultrasound-guided transversalis fascial plane block
  Interventions: Other: Transversalis Fascial Plane Block
- Quadratus Lumborum Block Group (Active Comparator): Patients will receive ultrasound-guided quadratus lumborum block
  Interventions: Other: Quadratus Lumborum Plane Block

INTERVENTIONS:
Other: Transversalis Fascial Plane Block — Patients will receive ultrasound-guided transversalis fascial plane block with 0,3 ml/kg of bupivacaine 0.25% just after general anesthesia induction
  Other Names: TFPB
  Arms: Transversalis Fascial Plane Block Group
Other: Quadratus Lumborum Plane Block — Patients will receive ultrasound-guided quadratus lumborum plane block with 0,3 ml/kg of bupivacaine 0.25% just after general anesthesia induction
  Other Names: QLB III
  Arms: Quadratus Lumborum Block Group

SUMMARY:
Regional anesthetic techniques; they reduce postoperative morbidity, provide early mobilization and provide great advantages by significantly reducing the need for narcotic analgesics. Regional anesthetic techniques are widely used in our clinic for postoperative analgesia, especially in infants and children. In patients undergoing lower abdominal surgery, postoperative analgesia is usually provided by systemic opioids and neuraxial methods. Complications such as sedation, respiratory depression, itching, nausea, vomiting and possible paraplegia or bleeding of neuraxial methods due to the use of opioids seem to be the biggest disadvantages of these two methods. Transversalis fascial plane (TFP) block is a regional anesthesia technique that provides intraoperative and postoperative analgesia as an alternative to caudal and epidural analgesia, especially in children. Transversalis fascial plane (TFP) block was first described in 2009. TFP block has been shown to be effective as an alternative to epidural analgesia and as part of a multimodal postoperative analgesic approach in lower abdominal and pelvic surgeries in children. Quadratus lumborum block (QLB) is a widely used regional anesthesia technique. It is used in pediatric patients to reduce postoperative pain in supraumbilical or infraumbilical surgeries. As a common result of all approaches, the main effect in quadratus lumborum block is anesthesia of the lateral cutaneous branches. In our center, the investigators have been using both methods, alone or in combination, routinely for a long time, and the investigators aim to compare the two methods in this study. This study consists of comparing two domain blocks known as part of multimodal analgesia.

DETAILED DESCRIPTION:
Transversalis fascial plane block and quadratus lumborum block are performed under general anesthesia just before the surgical incision, unless there are contraindications for the procedure for every patient scheduled for elective infraumbilical surgery in our center. In our study, patients will be divided into 2 groups and the effectiveness of trunk plan blocks, which are part of multimodal analgesia, will be compared. In the first group there will be patients who underwent transversalis fascial plane block (TFPB) alone, and in the second group there will be patients who underwent type III quadratus lumborum block (QLB). Post-operative pain scores with the Face, Leg, Activity, Cry, Consolability (FLACC) score will be recorded in 2-6-12-24th hours. Between both groups, postoperative analgesia need, time of analgesia need, presence of nausea and vomiting, surgeon and parent satisfaction will be followed up and recorded. All patients are operated under general anesthesia. General anesthesia is maintained with inhalation anesthesia. At the end of the surgery, the patient is awakened and taken to the recovery unit. In this prospective randomized study, the investigators will compare the efficacy of these two blocks, which are part of multimodal analgesia, with postoperative analgesic consumption. Postoperative patient comfort, complications, demographic findings will be used as data.

ELIGIBILITY:
Inclusion Criteria:

* Parental acceptation to participate and signed written consent
* Aged between 3 and 7
* American Society of Anesthesiologists (ASA) physical score I or II
* Elective infra umbilical surgery

Exclusion Criteria:

* Parental refusal to participate
* Known allergy to local anesthetics
* American Society of Anesthesiologists (ASA) physical score ≥ III
* Coagulopathy
* Hypersensitivity history to the agents to be used
* Local infections
* Known anatomically or systemic disorder
* Known growth and developmental retardation

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
Total dose of paracetamol consumption | in the first 24 hour postoperatively
  Total dose of paracetamol consumption in the ward

SECONDARY OUTCOMES:
FLACC score | in the first 24 hour postoperatively
  Postoperative FLACC score in the ward. FLACC score is a 10 point behavioral face, leg, activity, cry, consolability pain scale with a minimum score of 0 and a maximum of 10.
The 1st time to rescue analgesic need | in the first 24 hour postoperatively
  The time to ask for postoperative analgesia is the time from the end of operation to patient reporting FLACC score ≥ 4.
Number of postoperative nausea and vomiting | in the first 24 hour postoperatively
  Postoperative nausea and vomiting presence
Parental satisfaction level | in the first 24 hour postoperatively
  Parental satisfaction level will be evaluated using a five-point Likert scale 5= very satisfied 4= satisfied 3= neutral 2= dissatisfied
  1= very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Onur Baran, Asst. Prof., Study Chair — Namik Kemal University; Ayhan Şahin, Asst. Prof., Principal Investigator — Namik Kemal University; Cavidan Arar, Prof., Study Director — Namik Kemal University
Locations (1):
- Tekirdag Namik Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelbaser I, Mageed NA, El-Emam EM, ALseoudy MM, Elmorsy MM. Preemptive analgesic efficacy of ultrasound-guided transversalis fascia plane block in children undergoing inguinal herniorrhaphy: a randomized, double-blind, controlled study. Korean J Anesthesiol. 2021 Aug;74(4):325-332. doi: 10.4097/kja.20601. Epub 2020 Dec 14. PMID 33307633
- [Background] Arafa SK, Elsayed AA, Hagras AM, Shama AAA. Pediatric Postoperative Pain Control With Quadratus Lumborum Block and Dexamethasone in Two Routes With Bupivacaine: A Prospective Randomized Controlled Clinical Trial. Pain Physician. 2022 Oct;25(7):E987-E998. PMID 36288584
- [Background] Black ND, Malhas L, Jin R, Bhatia A, Chan VWS, Chin KJ. The analgesic efficacy of the transversalis fascia plane block in iliac crest bone graft harvesting: a randomized controlled trial. Korean J Anesthesiol. 2019 Aug;72(4):336-343. doi: 10.4097/kja.d.18.00352. Epub 2019 Mar 19. PMID 30886131
- [Background] Ahiskalioglu A, Aydin ME, Doymus O, Yayik AM, Celik EC. Ultrasound guided transversalis fascia plane block for lower abdominal surgery: First pediatric report. J Clin Anesth. 2019 Aug;55:130-131. doi: 10.1016/j.jclinane.2018.12.046. Epub 2019 Jan 15. No abstract available. PMID 30658324
- [Background] Chakraborty A, Goswami J, Patro V. Ultrasound-guided continuous quadratus lumborum block for postoperative analgesia in a pediatric patient. A A Case Rep. 2015 Feb 1;4(3):34-6. doi: 10.1213/XAA.0000000000000090. PMID 25642956